CLINICAL TRIAL: NCT03292666
Title: The Comparative Effectiveness of Warfarin and New Oral Anticoagulants for the Extended Treatment of Venous Thromboembolism
Brief Title: Anticoagulation Length of ThErapy and Risk of New Adverse evenTs In Venous thromboEmbolism Study
Acronym: ALTERNATIVE
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NOACs-1510-32651
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Venous Thromboembolism; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Venous Thromboembolism; Hemostatic Disorders | interventions — Anticoagulants; Warfarin; Dabigatran; Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extended anticoagulation: Patients with acute VTE treated with oral anticoagulants for > 3 months
  Interventions: Drug: Oral Anticoagulant
- No extended anticoagulation: Patients with acute VTE treated with oral anticoagulants for no longer than 3 months

INTERVENTIONS:
Drug: Oral Anticoagulant — Oral anticoagulants used to treat or prevent venous thromboembolism
  Other Names: warfarin, dabigatran, rivaroxaban, apixaban, edoxaban
  Groups: Extended anticoagulation

SUMMARY:
The proposed research seeks to provide insights on the contemporary epidemiology, treatment, and outcomes of VTE, including examining the uptake of new treatment strategies, the efficacy and safety of different anticoagulant options, and the impact of venous thromboembolism on patient-defined outcomes, such as quality-of-life, symptom burden, and treatment satisfaction. This information is crucial to helping clinicians and patients choose between various treatment options for venous thromboembolism in order to achieve the best possible balance between the risks, benefits, and impact on health.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a leading cause of cardiovascular death and continues to be a major public health issue in the United States. The cornerstone of current VTE treatment is anticoagulation, typically given for ≥ 3 months during the acute phase of thrombosis. Afterwards, extended-duration anticoagulation can be considered for selected higher-risk patients. Treatment options for VTE have expanded substantially in recent years, most notably through the availability of direct oral anticoagulants (DOACs). Yet there are many remaining gaps in the understanding of how to manage VTE to maximize net clinical benefit.

The long-range objective of this project is to reduce the morbidity and mortality associated with VTE in adults and evaluate contemporary treatment patterns and long-term outcomes after VTE. This initial phase of the study will assemble an observational cohort of adults with VTE diagnosed between 2010-2018. Study subjects will be identified from two integrated healthcare delivery systems (Kaiser Permanente Northern California and Kaiser Permanente Southern California) and followed until December, 2019. Data will be obtained from administrative and electronic health records, supplemented with a cross-sectional patient survey.

The first two aims will be to compare the rates of recurrent VTE and hemorrhage between (1) extended anticoagulation vs. no extended anticoagulation after VTE; and (2) DOAC vs. warfarin treatment of VTE. The third specific aim is to describe patient-defined outcomes in adults with VTE in the current treatment era. This will be accomplished by surveying subjects with VTE to collect data on generic and disease-specific quality-of-life as well as on anticoagulant treatment satisfaction. Combining clinical, outcome, and survey data with administrative data will create a contemporary cohort of VTE patients that can serve as a rich source of information for use in facilitating comparative effectiveness research addressing optimal VTE management within real-world practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years) enrolled in Kaiser Permanente Northern California or Kaiser Permanente Southern California
* Index VTE event, defined as an incident clinical encounter (inpatient, emergency department, or outpatient) with a primary or secondary diagnosis of VTE during the time period January 1, 2010 to December 31, 2018
* Anticoagulant prescription (oral or parenteral) filled after index VTE discharge/encounter date
* Continuous outpatient anticoagulant therapy for ≥ 3 months from fill date of prescription
* Continuous pharmacy benefits and health plan membership for at least 12 months before the index VTE event date

Exclusion Criteria:

- Incomplete information on age and sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source populations for the study will be adults diagnosed with acute venous thromboembolism who were enrolled in Kaiser Permanente Northern California or Kaiser Permanente Southern California, two large, integrated healthcare delivery systems in California.
Sampling Method: Non-Probability Sample
Enrollment: 39603 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism | From the index VTE date until death, disenrollment from the health system, or the end of the planned outcome assessment (December 31, 2019)
  Recurrent VTE will be defined as a new VTE encounter that is occurs after the index VTE event date. The encounter must represent a new diagnosis or symptomatology that is attributable to VTE.
Hospitalization for hemorrhage | From the index VTE date until death, disenrollment from the health system, or the end of the planned outcome assessment (December 31, 2019)
  Hospitalization for extracranial or intracranial hemorrhage

SECONDARY OUTCOMES:
Death | From the index VTE date until disenrollment from the health system or the end of the planned outcome assessment (December 31, 2019)
  All-cause death
Health-related quality of life | years 2018 and 2019
  Generic health-related quality of life, measured according to the 36 item Short Form Survey
Anticoagulant treatment satisfaction | years 2018 and 2019
  Anti-Clot Treatment Satisfaction Scale

CONTACTS AND LOCATIONS:
Overall Officials: Margaret C. Fang, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Oakland, California
  - Kaiser Permanente Southern California, Pasadena, California

IPD SHARING:
Plan to Share IPD: No